CLINICAL TRIAL: NCT02363985
Title: Using Stable Isotope Techniques to Monitor and Assess the Vitamin A Status of Children Susceptible to Infection in Ethiopia
Brief Title: Using Stable Isotope Techniques to Monitor and Assess the Vitamin A Status of Children Susceptible to Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ethiopian Public Health Institute (Other Government)
Collaborators: International Atomic Energy Agency (Other Government)
Responsible Party: Principal Investigator, Tesfaye Hailu, Researcher, Ethiopian Public Health Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: EPHI_IAEA_P6047
Record Dates: First submitted 2015-02-10; First posted 2015-02-16 (Estimated); Last update posted 2017-12-12 (Actual); Status verified 2017-12

CONDITIONS: Vitamin A Deficiency
MeSH Terms: conditions — Vitamin A Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multiple vitamin A exposer (Other): 55 children who are using
  * Mega-dose vitamin A supplementation
  * Food diversification (promotion and education on vitamin A rich food consumption)
  * Promotion of orange flash sweet potato production and consumption in collaboration with international potato center (CIP) in one of the study area
  Interventions: Dietary Supplement: Mega-dose of vitamin A supplement
- Only vitamin A supplementation (Other): 55 children who are using
  * Mega-dose vitamin A supplementation
  * Food diversification (promotion and education on vitamin A rich food consumption)
  Interventions: Dietary Supplement: Mega-dose of vitamin A supplement

INTERVENTIONS:
Dietary Supplement: Mega-dose of vitamin A supplement — vitamin A supplementation normally given every six months for under five children in Ethiopia. In addition, there is also dietary intervention like orange flash sweet potato and promotion of other vitamin A rich foods to tackle vitamin A deficiency in Ethiopia.

SUMMARY:
The combination of infectious diseases and malnutrition is the most prevalent, preventable public health problem in the world, responsible for millions of deaths annually, particularly in infants and children. Approximately 13 million children die each year in developing countries from infectious diseases, with the majority of these deaths related to malnutrition. The relationship between infections and malnutrition is synergistic, each further compromising the outcome of the other. Malnutrition compromises natural immunity leading to increased susceptibility to infections, more frequent and prolonged disease episodes, and increased severity of disease. Likewise, infections can aggravate or precipitate malnutrition through decreased appetite and food intake, nutrient malabsorption, nutrient loss or increased metabolic needs. Another issue is that infections (as well as overweight and obesity status) affect nutritional biomarkers making it difficult to assess the real magnitude of some nutritional problems. This is the case of vitamin A. Vitamin A deficiency is defined to be of severe public health importance if 20% or more of a defined population has a serum retinol concentration of less than 0.7 µmol/L. However, circulating concentrations of serum retinol are reduced by infections and in such situations serum retinol concentration is not a good indicator of vitamin A status. Serum acute-phase proteins can indicate the severity and duration of an infection. Correcting vitamin A deficiency is addressed in Ethiopia through vitamin A supplementation of children, dietary diversity and using bio-fortified foods. However, assessing vitamin A status, and the effectiveness of government interventions, is challenging in settings where infectious diseases are endemic, as in most area of the country. Evaluation of vitamin A status is relatively insensitive when based on changes in serum retinol concentrations, which are homeostatically controlled and negatively affected by subclinical infections. Liver stores of vitamin A, the best indicator of vitamin A status, cannot be routinely evaluated. The isotope dilution technique is the preferred method for determining vitamin A status and assessing the efficacy and effectiveness of intervention programs aimed at improving vitamin A status. It is the only indirect assessment method that provides a quantitative estimate of vitamin A status across the continuum of deficient to excessive stores.

DETAILED DESCRIPTION:
Vitamin A deficiency is the leading cause of preventable blindness in children and is associated with a higher risk of under five mortality. Approximately 250,000 to 500,000 children in developing countries become blind each year owing to vitamin A deficiency, with the highest prevalence in South Asia and Africa. In Africa, many countries have implemented vitamin A interventions of mega-dose supplementation for children under 5 years, sometimes in combination with food fortification programs.

Vitamin A deficiency is a major nutritional concern; with more than 37.7% of under five children being vitamin A deficient by serum retinol and 50.7% had been sick in the previous 15 days in Ethiopia. Vitamin A deficiency is addressed in the country through vitamin A supplementation every six months for 6-59 months of children and during the first 45 days of delivery for lactating mothers. There are also other vitamin A intervention programs like bio-fortification of orange flesh sweet potato (OFSP) in pocket areas. Unfortunately, assessing vitamin A status, and the effectiveness of government interventions, is challenging in settings where infectious diseases are endemic, as in most African countries including Ethiopia. This is because serum retinol concentration decreases during infection due to the acute phase response.

The overall national prevalence of any helminthes infection in Ethiopia was 29.8% with variable degree of prevalence among regions, where by southern nation nationality people (SNNP) (51%) and Gambella (51%) have the highest prevalence. A survey in 13 foods for education program-supported schools in the SNNP region indicated that prevalence of soil transmitted helminthiasis infections are 44.4%. The proportion of school children infected with any parasite species was 55.4%. A. lumbricoides was the most prevalent species 32.1%, followed by hookworm 21.7%.

Forty seven subjects (26 male and 21 female) met the survey definition of smear positive tuberculosis (TB) cases, with a prevalence of 108/100,000 (72-138). From smear positive TB cases, 37(78.7%) were new cases, 2(4.3%) were on treatment, and 8(17%) were previously treated in the last five years. Malaria prevalence is 4.5% in the malaria endemic area.

Evaluation of Vitamin A status is relatively insensitive when based on changes in serum retinol, which is homeostatically controlled and negatively affected by subclinical infections. Liver stores of vitamin A are the best indicator of vitamin A status, but cannot be routinely evaluated. The isotope dilution technique is the preferred method for determining vitamin A status and assessing the efficiency and effectiveness of intervention programs. It is the only indirect assessment method that provides a quantitative estimate of vitamin A status across the continuum from deficient to excessive vitamin A.

Hence, this project will assess the vitamin A and inflammatory status of 3-5 year old children 4-5 months after their semi-annual mega-dose vitamin A supplementation. The results will indicate the proportions of sampled children with low, normal or high vitamin A status, how inflammation (from obesity or recent infection or injury) affects assessment of vitamin A status using different vitamin A assessment methods, and how status differs by country, in possible association with food fortification practices.

Gap /Problem /Needs Analysis

The combination of infectious diseases and malnutrition is the most prevalent, preventable public health problem in the world, responsible for millions of deaths annually, particularly in infants and children. Approximately 13 million children die each year in developing countries from infectious diseases, with the majority of these deaths related to malnutrition. The relationship between infections and malnutrition is synergistic, each further compromising the outcome of the other. Malnutrition compromises natural immunity leading to increased susceptibility to infections, more frequent and prolonged disease episodes, and increased severity of disease. Likewise, infections can aggravate or precipitate malnutrition through decreased appetite and food intake, nutrient mal-absorption, nutrient loss or increased metabolic needs. Severe malnutrition often masks symptoms and signs of infectious diseases making prompt clinical diagnosis and treatment very difficult. Another issue is that infections (as well as overweight and obesity status) affect nutritional biomarkers making it difficult to assess the real magnitude of some nutritional problems. This is the case of vitamin A. Vitamin A deficiency is defined to be of severe public health importance if 20% or more of a defined population has a serum retinol concentration of less than 0.7 µmol/L. However, circulating concentrations of serum retinol are reduced by infections and in such situations serum retinol concentration is not a good indicator of vitamin A status. Infections are accompanied by an acute phase response, and serum acute-phase proteins can indicate the severity and duration of an infection. Acute-phase proteins, such as C-reactive protein (CRP), increase within the first 6h of infection, and reach their maximum concentrations within 24-48h. However, α1-acid-glycoprotein (AGP) rises more slowly, with maximum concentrations 2-5 days after infection. Vitamin A deficiency is a major nutritional concern in poor societies affecting 190 million children globally.

Vitamin A is an essential nutrient needed for the visual system, and maintenance of cell function for growth, epithelial integrity, red blood cell production, immunity and reproduction. All infants are born with low stores and depend on vitamin A from breast milk to initially accumulate and maintain adequate stores. Infants of vitamin A depleted women are at greater risk of becoming vitamin A deficient early in life, especially if they are not breast fed. Correcting vitamin A deficiency is addressed by some African countries through vitamin A supplementation of children and food fortification programs. However, assessing vitamin A status, and the effectiveness of government interventions, is challenging in settings where infectious diseases are endemic, as in most African countries. Evaluation of vitamin A status is relatively insensitive when based on changes in serum retinol concentrations, which are homeostatically controlled and negatively affected by subclinical infections. Liver stores of vitamin A, the best indicator of vitamin A status, cannot be routinely evaluated. The isotope dilution technique is the preferred method for determining vitamin A status and assessing the efficacy and effectiveness of intervention programs aimed at improving vitamin A status. It is the only indirect assessment method that provides a quantitative estimate of vitamin A status across the continuum of deficient to excessive stores. Thus, this technique can be used for assessing vitamin A status in populations at risk of excessive status due to exposure to too much vitamin A through combined supplementation and consumption of fortified foods and/or preformed vitamin A-rich foods. The aim of this project is to use nuclear techniques to evaluate vitamin A nutritional status of young children during semi-annual administration of vitamin A supplements, and to assess how this relates to infection status.

The International Atomic Energy Agency (IAEA) has provided significant support on use of stable isotopes in assessing body composition and breast milk to Member States in Africa, it is now establishing the stable isotope technique to assess vitamin A body stores in Cameroon and Zambia (and additional implementation is possible in other country) for use throughout the region. These inputs will be used in this project to provide key information to stakeholders on how vitamin A intervention programs affect vitamin A status in children and how infections affect vitamin A status or validity of stable isotope techniques.

Role of nuclear technology The nuclear techniques used will be the deuterated- and 13 Carbon-retinol body pool measurements to assess vitamin A status. These nuclear methods are useful across the continuum of nutritional status from deficient to adequate to excess, in contrast with the more common measurement of serum retinol concentrations. In addition, the presence of infection/inflammation is less likely to interfere with interpretation of the nuclear method than that of the serum retinol method, but this will be investigated in this series of studies. This method is already being established in 2-3 countries and the serum retinol method is established in approximately 8 countries. Further use of the deuterated retinol body pool size nuclear method will contribute to capacity building in Africa, where vitamin A supplementation of children and widespread fortification are routine. The combination of multiple vitamin A interventions requires continuous monitoring. The IAEA is expected to provide technical and logistical support for the use of isotope dilution methods and facilitate Fellowships, Training, Scientific Visits, Expert Missions and Supplies.

ELIGIBILITY:
Inclusion Criteria:

* 3-5 years, planning to move from the study area for the duration of the study, and do not have severe illness at the time of enrollment.

Exclusion Criteria:

* severe anaemia, severe acute malnutrition, obesity or clinically defined severe illness, such as dehydration, severe diarrhoea or severe respiratory illness.

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 138 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Total body pool size vitamin A (µmol) | within the coming 2 years
  estimate the total body pool size vitamin A in preschool child in Ethiopia using stable isotope technique
Liver Vitamin A store (µmol/g) | within the coming 2 years
  Liver Vit A store (µmol/g) cut off <= 0.07
Serum retinol (µmol/l) | within the coming 2 years
  Serum retinol (µmol/l) cut off <= 0.7

SECONDARY OUTCOMES:
level of infection | within the coming 2 years
  AGP and CRP
dietary intake | within the coming 2 years
  mean intake of beta carotene and dietary diversity score using 24 hour dietary recall
Anthropometry measurement | within the coming 2 years
  Weight for Height Z-score, Weight for Age Z-score, Height for Age Z-score and middle upper arm circumference
socioeconomic status | within the coming 2 years
  household (HH) family size, marital status of the mother, head of the HH, source of drinking wate, highest level of education the head of HH attend
Morbidity | within the coming 2 years
  medical history of the child enrolled in the study such as diarrhea, cough, fever, malaria, rashes, measles, vaccination, vitamin A supplementation, durg for intestinal deworming, iron supplementation.

CONTACTS AND LOCATIONS:
Overall Officials: Cornelia Loechl, PhD, Study Director — International Atomic Energy Agency
Locations (1):
- Ethiopian Public Health Institute, Addis Ababa, Ethiopia